CLINICAL TRIAL: NCT03392207
Title: Active Surveillance for Adverse Events Following Immunization With the Trivalent Influenza Vaccine (2018 Southern Hemisphere Season) Produced at Butantan Institute
Brief Title: Active Surveillance for Adverse Events Following Immunization With the Butantan Trivalent Influenza Vaccine (2018)
Acronym: FLU-06-IB
Status: Completed | Type: Observational
Sponsor: Butantan Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: FLU-06-IB
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Respiratory Tract Infections; Virus Diseases; Vaccines; Physiological Effects of Drugs
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Care Professionals: Health care professionals receiving the seasonal influenza vaccine (2018) produced by Butantan Institute.
  Interventions: Biological: Seasonal Influenza Vaccine
- Elderly: Elderly (age 60 or more) receiving the seasonal influenza vaccine (2018) produced by Butantan Institute.
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — Trivalent, Fragmented, Inactivated Seasonal Influenza Vaccine (2018 Southern Hemisphere Season) produced at Butantan Institute

SUMMARY:
Rationale and Background: Since 2013, Butantan Institute has been performing passive pharmacovigilance activities related to its triavalent, fragmented and inactivated vaccine (IB TIV).

Objetive: To conduct an active surveillance study focusing on the elderly and health care professionals as part of Butantan pharmacovigilance plan, while passive surveillance activities will continue. The pharmacovigilance plan, via active surveillance, is being implemented in response to WHO requirements for pre-qualification of IB TIV.

DETAILED DESCRIPTION:
Study Design: This is a prospective cohort study. Population: Target groups for vaccination defined by The National Immunization Program of Brazil: healthcare workers and elderly (people over 60 years old). Study Size: A total of 400 individuals (150 health care workers and 250 elderly), presenting for immunization with IB TIV, and who agree to participate after providing Informed Consent.

ELIGIBILITY:
Inclusion Criteria:

* Health Care Professional; or
* Elderly (age 60 or more); and
* To have indication to be vaccinated against influenza, according the the Brazilian National Immunazition Programme; and
* To be available to participate in the study throughout its duration (6 weeks after any vaccine dose administered); and
* To demonstrates interest to participate in the study as registered in the informed consent form (ICF).

Exclusion Criteria:

* Known systemic hypersensitivity to eggs or to any component of the vaccine;
* Suspected or confirmed fever in the 3 days prior to vaccination or axillary temperature greater than 37.8 ° C on the day of vaccination;
* History of severe adverse reaction after previous administration of an Influenza vaccine within 6 weeks following vaccination;
* History of Guillain-Barre Syndrome or other demyelinating disease;
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
* Any other condition in the opinion of the investigator that justifies exclusion from participation.

Ages: 18 Years to 130 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People eligible for immunization with seasonal influenza vaccine, focusing on: elderly and health care workers.
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
number of participants with adverse events following immunization (AEFI), 42 days post-vaccination. | 42 days post-vaccination
  to estimate the incidence of AEFI associated with administration of the trivalent, fragmented, inactivated influenza vaccine (2018 Southern Hemisphere Season) produced at Butantan Institute within 42 days post-vaccination.

SECONDARY OUTCOMES:
number of solicited AEFI, 14 days post-vaccination. | 14 days post-vaccination
  to estimate the incidence of solicited AEFI associated with administration of the trivalent, fragmented, inactivated influenza vaccine (2018 Southern Hemisphere Season) produced at Butantan Institute within 14 days post-vaccination.
number of unsolicited AEFI, 14 days post-vaccination. | 14 days post-vaccination
  to estimate the incidence of unsolicited adverse events following immunization (AEFI) associated with administration of the trivalent, fragmented, inactivated influenza vaccine (2018 Southern Hemisphere Season) produced at Butantan Institute within 14 days post-vaccination.
number of unsolicited AEFI, 42 days post-vaccination. | 42 days post-vaccination
  to estimate the incidence of unsolicited adverse events following immunization (AEFI) associated with administration of the trivalent, fragmented, inactivated influenza vaccine (2018 Southern Hemisphere Season) produced at Butantan Institute within 42 days post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Precioso, MD, PhD, Study Director — Instituto Butantan
Locations (2):
- Brazil (2):
  - Crie - Unifesp, São Paulo, São Paulo
  - Avenida Vital Brasil 1500, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided